CLINICAL TRIAL: NCT00107419
Title: Phase II Trial of Pemetrexed for Advanced Chondrosarcomas
Brief Title: S0423 Pemetrexed Disodium in Treating Patients With Recurrent and Unresectable or Metastatic Chondrosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000415848; S0423 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Sarcoma
Keywords: chondrosarcoma
MeSH Terms: conditions — Sarcoma; Chondrosarcoma | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pemetrexed (Experimental): pemetrexed
  Interventions: Drug: pemetrexed disodium

INTERVENTIONS:
Drug: pemetrexed disodium — pemetrexed, 500 mg/m2, IV, every 21 days until two cycles after complete response or until progression

SUMMARY:
RATIONALE: Pemetrexed disodium may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well pemetrexed disodium works in treating patients with recurrent and unresectable or metastatic chondrosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate (confirmed and unconfirmed complete response and partial response) in patients with recurrent and unresectable or metastatic chondrosarcoma treated with pemetrexed disodium.

Secondary

* Determine the toxicity of this drug in these patients.
* Correlate, preliminarily, response rates with deletions of methylthioadenosine phosphorylase (MTAP), as analyzed by fluorescence in-situ hybridization (FISH), in patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to prior chemotherapy (yes vs no).

Patients receive pemetrexed disodium IV over 10 minutes on day 1. Courses repeat every 21 days* in the absence of disease progression or unacceptable toxicity. Beginning 7 days before the first dose of pemetrexed disodium and continuing until 21 days after the completion of pemetrexed disodium, patients receive cyanocobalamin (vitamin B_12) intramuscularly once every 63 days and oral folic acid once daily.

NOTE: *The duration of course 1 is 28 days; the duration of all subsequent courses is 21 days.

Patients achieving a complete response (CR) receive 2 additional courses beyond CR. Patients achieving a confirmed partial response (PR) that is resectable, proceed to surgical resection and then receive 2 additional courses of therapy after recovering from surgery. Patients achieving a confirmed PR that is not resectable continue treatment in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months until disease progression and then every 6 months for up to 5 years.

PROJECTED ACCRUAL: A total of 40-75 patients (20-40 in the previously treated stratum and 20-35 in the previously untreated stratum) will be accrued for this study within 20-37.5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed chondrosarcoma

  * Histologic grade G2 or G3
  * Recurrent and unresectable OR metastatic disease
* Measurable disease by x-ray, scan, ultrasound, or physical examination
* No known CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin < 1.5 times upper limit of normal (ULN)
* SGOT or SGPT < 2.5 times ULN (5 times ULN if liver metastases are present)

Renal

* Creatinine clearance > 45 mL/min

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Able to swallow oral medication
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 28 days since prior biologic therapy for this malignancy

Chemotherapy

* More than 28 days since prior chemotherapy for this malignancy

Endocrine therapy

* Not specified

Radiotherapy

* At least 60 days since prior radiotherapy to the target lesion*
* No concurrent radiotherapy NOTE: *Target lesion must have demonstrated disease progression after completion of therapy

Surgery

* At least 21 days since prior surgery and recovered

Other

* More than 28 days since prior investigational drugs for this malignancy
* At least 60 days since prior embolization or radiofrequency ablation to the target lesion*
* No more than 2 prior treatment regimens for this malignancy
* No concurrent antiretroviral therapy for HIV-positive patients NOTE: *Target lesion must have demonstrated disease progression after completion of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-09; Primary Completion 2007-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Response rate as measured by RECIST criteria | every 9 weeks during treatment
  x-rays or scans

SECONDARY OUTCOMES:
Toxicity as measured by CTC v 3.0 | every 3 weeks during treatment
  side-effect evaluation
Response rate compared with methylthioadenosine phosphorylase (MTAP) deletions as measured by fluorescence in-situ hybridization (FISH) retrospectively | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Warren A. Chow, MD, Study Chair — City of Hope Comprehensive Cancer Center; Ernest C. Borden, MD, Study Chair — The Cleveland Clinic; Vivien H.C. Bramwell, MB, BS, PhD, FRCP, Study Chair — Tom Baker Cancer Centre - Calgary; George D. Demetri, MD, Study Chair — Dana-Farber Cancer Institute; Margaret von Mehren, MD, Study Chair — Fox Chase Cancer Center
Locations (58):
- United States (58):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Oregon Health & Science University Cancer Institute, Portland, Oregon
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Medical City Dallas Hospital, Dallas, Texas
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming